CLINICAL TRIAL: NCT02002234
Title: Hemicraniectomy for Malignant Middle Cerebral Artery Infarction (HeMMI): A Single Center Randomized Controlled Clinical Trial
Brief Title: Hemicraniectomy for Malignant Middle Cerebral Artery Infarction (HeMMI)
Acronym: HeMMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment for the study was terminated due to slow recruitment
Sponsor: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIDO 2002
Record Dates: First submitted 2013-11-07; First posted 2013-12-05 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2014-02

CONDITIONS: Infarction
Keywords: Hemicraniectomy, stroke, decompressive surgery, HeMMI
MeSH Terms: conditions — Infarction; Stroke

ARMS (2):
- Medical Treatment Arm (Other): Received standardized medical therapy in an intensive care unit (ICU), which included elevation of the head of bed at 30°, intermittent hyperventilation administered, and intravenous mannitol. Mean arterial pressure was maintained above 90 mm Hg. Hemoglobin concentration was maintained at all times above 90 g/L. Hyperglycemia, hyperthermia and hypotension were avoided or corrected when present.
  Interventions: Procedure: Standard medical treatment
- Surgery with Medical Treatment Arm (Other): Aside from receiving standardized medical therapy, decompressive hemicraniectomy was performed by removing a large bone flap at least 12 cm in diameter and included parts of the frontal, temporal, parietal and occipital bones, with further craniectomy to the floor of the temporal fossa. The dura was opened widely and duraplasty was performed using periosteum and temporalis fascia. The bone flap was either stored in a subcutaneous pocket in the abdomen or placed in the bone bank. Cranioplasty was performed during a separate admission on an elective basis not earlier than 6 months from the initial surgery.
  Interventions: Procedure: Hemicraniotomy

INTERVENTIONS:
Procedure: Hemicraniotomy — Hemicraniotomy involves removing a large bone flap at least 12 cm in diameter and included parts of the frontal, temporal, parietal and occipital bones, with further craniectomy to the floor of the temporal fossa. The dura was opened widely and duraplasty was performed using periosteum and temporalis fascia. The bone flap was either stored in a subcutaneous pocket in the abdomen or placed in the bone bank.
  Arms: Surgery with Medical Treatment Arm
Procedure: Standard medical treatment — Standard medical treatment involves elevation of the head of bed at 30°, intermittent hyperventilation administered, and intravenous mannitol. Mean arterial pressure was maintained above 90 mm Hg. Hemoglobin concentration was maintained at all times above 90 g/L.
  Arms: Medical Treatment Arm

SUMMARY:
A single-centered, randomized, controlled clinical trial comparing standardized medical care alone with standardized medical care and decompressive hemicraniectomy to determine the effectiveness of decompressive surgery more definitively in patients with clinical signs of infarction of the Middle Carotid Artery (MCA) territory.

DETAILED DESCRIPTION:
A single-centered, randomized, controlled clinical trial comparing standardized medical care alone with standardized medical care and decompressive hemicraniectomy to determine the effectiveness of decompressive surgery more definitively in patients with clinical signs of infarction of the MCA territory and and who arrived at the hospital within 72 hours of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 65 years old who presented with clinical signs of infarction of the MCA territory and who arrived at the hospital within 72 hours of symptom onset. Other inclusion criteria included a Glasgow coma score (GCS) of 6 to14 in patients with right MCA infarction or GCS 5 to 9 in patients with left MCA infarction (adjusted to account for effect on speech deficit on GCS scores), or GCS of 15 on arrival but subsequently deteriorated neurologically as defined by a score of ≥1 on the level of consciousness item of the National Institutes of Health Stroke Scale (NIHSS);computed tomography (CT) scan of the head showing ischemic changes corresponding to more than 50% of the MCA territory with or without involvement of other vascular territories;and written informed consent from the patient or a legal representative.

Exclusion Criteria:

* Patients with previous disabling neurological disease, an estimated premorbid modified Rankin Scale (mRS) score >2; terminal illness; presence of serious medical comorbidities like end-stage renal failure and cardiac disease with severe hemodynamic compromise; infarction due to surgical complications or vasospasm; primary intracranial hemorrhage; coagulopathies; and high risk for surgery upon assessment by the medical team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Functional status measured by modified Rankin Score (mRS) | up to six months
  The primary outcome measure was functional status measured by the modified Rankin Score, dichotomized as a good status (mRS 0-3) or poor status (mRS 4-6). A score of mRS 0-3 indicates functional status ranging from no symptoms to "moderate disability" (defined in the modified Rankin Scale as requiring some help, but able to walk without assistance); mRS 4-6 indicates functional status ranging from "moderately severe disability" (unable to walk or to attend to own bodily needs without assistance) through to death. A cut off of mRS 3 was adopted a priori because the ability to walk independently, with or without the help of a device, was considered a favorable outcome. Follow-up assessments, including mRS, were at seven days, two weeks, one month, three months, and six months post-stroke.

SECONDARY OUTCOMES:
Survival measured by modified Rankin Score (mRS) | up to six months
  The Secondary outcome measure is the survival of the patients at six months measured using mRS scores dichotomized at mRS 0-4 and mRS 5-6 at six months. A score of mRS 0-4 indicates functional status ranging from no symptoms to "moderately severe disability" (unable to walk without assistance and unable to attend to own bodily needs without assistance); mRS 5-6 indicates functional status ranging from "severe disability" (bedridden, incontinent and requiring constant nursing care and attention) through to death. The latter outcome was considered because it was included in previous trial reports

CONTACTS AND LOCATIONS:
Overall Officials: Annabelle E Chua, MD, Principal Investigator — University of the Philippines Manila
Locations (1):
- Philippine General Hospital - University of the Philippines Manila, Manila, National Capital Region, Philippines